CLINICAL TRIAL: NCT03269929
Title: Comparison Between Music Therapy and Intravenous Midazolam 0,02 mg/kgBW in Reducing Preoperative Anxiety: Study on Patient Undergoing Brachytherapy With Spinal Anesthesia
Brief Title: Comparison Between Efficacy of Music Therapy and Intravenous Midazolam 0.02 mg/kgBW in Reducing Preoperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Christopher Kapuangan, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes018
Record Dates: First submitted 2017-07-19; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Music Therapy; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music therapy (Experimental)
  Interventions: Other: Music therapy
- Midazolam (Active Comparator)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Other: Music therapy — Subjects listened to music for 30 minutes before undergoing brachytherapy with spinal anesthesia
  Arms: Music therapy
Drug: Midazolam — Subjects received intravenous midazolam 0,02 mg/kgBW injection before undergoing brachytherapy with spinal anesthesia
  Arms: Midazolam

SUMMARY:
This study aimed to compare the efficacy of music therapy and midazolam 0,02 mg/kgBW in reducing preoperative anxiety on patients undergoing brachytherapy with spinal anesthesia

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study. Intravenous (IV) cannula had been set and The Amsterdam Preoperative Anxiety and Information (APAIS) score questionnaire was filled by the subject. Blood pressure, pulse rate, and mean arterial pressure were recorded. Subjects were then randomized into two groups (music therapy and midazolam). In music therapy group, subjects listened to music using headphone attached to music player for 30 minutes. Music player has been filled with variety of slow beat songs (60 - 80 BPM), including instrumental, pop, jazz, classical, and so forth. In midazolam group, subjects was given intravenous midazolam 0,02 mg/kgBW injection without listening to music. After injection, subjects are allowed to rest or sleep for 30 minutes. After intervention, APAIS score was filled by subjects with blood pressure, pulse rate, and mean arterial pressure recorded again. Subjects then were moved to brachytherapy room.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18-65 years old
* Undergoing one day care brachtherapy with spinal anesthesia
* American Society of Anesthesiologist (ASA) physical status of I-III
* Agreed to participate in this study and signed informed consent
* Able to read, write, and speak in Indonesian language.

Exclusion Criteria:

* Subjects with severe hearing impairment
* Subjects with cognitive/mental impairment based on medical record
* Subjects with previous routine use of antipsychotic and benzodiazepine drug
* Subjects with prior heart disease or uncontrolled hypertension.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
APAIS score | Day 1
Blood pressure | Day 1
Pulse rate | Day 1
Mean Arterial Pressure | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Central Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mohd Fahmi Z, Lai LL, Loh PS. Validation of the Malay version of the Amsterdam Preoperative Anxiety and Information Scale (APAIS). Med J Malaysia. 2015 Aug;70(4):243-8. PMID 26358022
- [Background] Caumo W, Schmidt AP, Schneider CN, Bergmann J, Iwamoto CW, Bandeira D, Ferreira MB. Risk factors for preoperative anxiety in adults. Acta Anaesthesiol Scand. 2001 Mar;45(3):298-307. doi: 10.1034/j.1399-6576.2001.045003298.x. PMID 11207465
- [Background] Hyde R, Bryden F, Asbury AJ. How would patients prefer to spend the waiting time before their operations? Anaesthesia. 1998 Feb;53(2):192-5. doi: 10.1046/j.1365-2044.1998.00268.x. PMID 9534647
- [Background] Bradt J, Dileo C, Shim M. Music interventions for preoperative anxiety. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD006908. doi: 10.1002/14651858.CD006908.pub2. PMID 23740695
- [Background] Wright KD, Stewart SH, Finley GA, Buffett-Jerrott SE. Prevention and intervention strategies to alleviate preoperative anxiety in children: a critical review. Behav Modif. 2007 Jan;31(1):52-79. doi: 10.1177/0145445506295055. PMID 17179531
- [Background] Griffin CE 3rd, Kaye AM, Bueno FR, Kaye AD. Benzodiazepine pharmacology and central nervous system-mediated effects. Ochsner J. 2013 Summer;13(2):214-23. PMID 23789008
- [Background] Sun GC, Hsu MC, Chia YY, Chen PY, Shaw FZ. Effects of age and gender on intravenous midazolam premedication: a randomized double-blind study. Br J Anaesth. 2008 Nov;101(5):632-9. doi: 10.1093/bja/aen251. Epub 2008 Sep 4. PMID 18772216
- [Background] Kain ZN, Sevarino F, Pincus S, Alexander GM, Wang SM, Ayoub C, Kosarussavadi B. Attenuation of the preoperative stress response with midazolam: effects on postoperative outcomes. Anesthesiology. 2000 Jul;93(1):141-7. doi: 10.1097/00000542-200007000-00024. PMID 10861157
- [Background] Marwick C. Music therapists chime in with data on medical results. JAMA. 2000 Feb 9;283(6):731-3. No abstract available. PMID 10683042
- [Background] Kamer S, Ozsaran Z, Celik O, Bildik O, Yalman D, Bolukbasi Y, Haydaroglu A. Evaluation of anxiety levels during intracavitary brachytherapy applications in women with gynecological malignancies. Eur J Gynaecol Oncol. 2007;28(2):121-4. PMID 17479673
- [Background] Wetsch WA, Pircher I, Lederer W, Kinzl JF, Traweger C, Heinz-Erian P, Benzer A. Preoperative stress and anxiety in day-care patients and inpatients undergoing fast-track surgery. Br J Anaesth. 2009 Aug;103(2):199-205. doi: 10.1093/bja/aep136. Epub 2009 May 30. PMID 19483203
- [Background] Mitchell M. Influence of gender and anaesthesia type on day surgery anxiety. J Adv Nurs. 2012 May;68(5):1014-25. doi: 10.1111/j.1365-2648.2011.05801.x. Epub 2011 Aug 2. PMID 21806671
- [Background] Cooke M, Chaboyer W, Schluter P, Hiratos M. The effect of music on preoperative anxiety in day surgery. J Adv Nurs. 2005 Oct;52(1):47-55. doi: 10.1111/j.1365-2648.2005.03563.x. PMID 16149980
- [Background] Bringman H, Giesecke K, Thorne A, Bringman S. Relaxing music as pre-medication before surgery: a randomised controlled trial. Acta Anaesthesiol Scand. 2009 Jul;53(6):759-64. doi: 10.1111/j.1399-6576.2009.01969.x. Epub 2009 Apr 14. PMID 19388893
- [Background] Leardi S, Pietroletti R, Angeloni G, Necozione S, Ranalletta G, Del Gusto B. Randomized clinical trial examining the effect of music therapy in stress response to day surgery. Br J Surg. 2007 Aug;94(8):943-7. doi: 10.1002/bjs.5914. PMID 17636513
- [Background] Bishop SJ. Neurocognitive mechanisms of anxiety: an integrative account. Trends Cogn Sci. 2007 Jul;11(7):307-16. doi: 10.1016/j.tics.2007.05.008. Epub 2007 Jun 5. PMID 17553730
- [Background] Nigussie S, Belachew T, Wolancho W. Predictors of preoperative anxiety among surgical patients in Jimma University Specialized Teaching Hospital, South Western Ethiopia. BMC Surg. 2014 Sep 5;14:67. doi: 10.1186/1471-2482-14-67. PMID 25189274
- [Background] Ploghaus A, Narain C, Beckmann CF, Clare S, Bantick S, Wise R, Matthews PM, Rawlins JN, Tracey I. Exacerbation of pain by anxiety is associated with activity in a hippocampal network. J Neurosci. 2001 Dec 15;21(24):9896-903. doi: 10.1523/JNEUROSCI.21-24-09896.2001. PMID 11739597
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Kupietzky A, Houpt MI. Midazolam: a review of its use for conscious sedation of children. Pediatr Dent. 1993 Jul-Aug;15(4):237-41. No abstract available. PMID 8247896
- [Background] Nordt SP, Clark RF. Midazolam: a review of therapeutic uses and toxicity. J Emerg Med. 1997 May-Jun;15(3):357-65. doi: 10.1016/s0736-4679(97)00022-x. PMID 9258787
- [Background] Golparvar M, Saghaei M, Sajedi P, Razavi SS. Paradoxical reaction following intravenous midazolam premedication in pediatric patients - a randomized placebo controlled trial of ketamine for rapid tranquilization. Paediatr Anaesth. 2004 Nov;14(11):924-30. doi: 10.1111/j.1460-9592.2004.01349.x. PMID 15500492
- [Background] Dundee JW, Halliday NJ, Harper KW, Brogden RN. Midazolam. A review of its pharmacological properties and therapeutic use. Drugs. 1984 Dec;28(6):519-43. doi: 10.2165/00003495-198428060-00002. PMID 6394264
- [Background] Kemper KJ, Danhauer SC. Music as therapy. South Med J. 2005 Mar;98(3):282-8. doi: 10.1097/01.SMJ.0000154773.11986.39. PMID 15813154
- [Background] Yinger OS, Gooding L. Music therapy and music medicine for children and adolescents. Child Adolesc Psychiatr Clin N Am. 2014 Jul;23(3):535-53. doi: 10.1016/j.chc.2013.03.003. Epub 2013 May 17. PMID 24975624
- [Background] Nilsson U. The anxiety- and pain-reducing effects of music interventions: a systematic review. AORN J. 2008 Apr;87(4):780-807. doi: 10.1016/j.aorn.2007.09.013. PMID 18395022
- [Background] Wang SM, Kulkarni L, Dolev J, Kain ZN. Music and preoperative anxiety: a randomized, controlled study. Anesth Analg. 2002 Jun;94(6):1489-94, table of contents. doi: 10.1097/00000539-200206000-00021. PMID 12032013